CLINICAL TRIAL: NCT05801367
Title: Allium Sativum Oil as Alternative Non-vital Pulpotomy Medicament in Primary Teeth- A Randomized Controlled Trial
Brief Title: Allium Sativum Oil as Alternative Non-vital Pulpotomy Medicament in Primary Teeth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Collaborators: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Mashal Mazhar, Dental Surgeon (Ex-Postgraduate trainee), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversityUHS
Record Dates: First submitted 2023-02-28; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Non-Vital Tooth
MeSH Terms: conditions — Tooth, Nonvital | interventions — formocresol; allyl sulfide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and assessors involved in the study from randomization, allocation, bacteriological outcome, and data analysis will be blinded to which medicament group the patients belonged as all data will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formocresol (Control-Gold standard-Group A) (Active Comparator): Premade Formocresol (Tricresol & Formalin) will be used in this research. Composition was Tricresol 35%, Formaldehyde (40%) 19%, excipient additive 100% (PD, Switzerland, ISO9001/ISO9001_2000/ ISO13485/CE_MARK), (Universal Dental Pvt, Ltd)
  Interventions: Drug: Formocresol
- Allium sativum oil (Experimental-Group B) (Experimental): Premade Allium sativum oil (Garlic oil) (Mohammad and Baroudi, 2015b) will be used in this research (SAC group of companies-9001:2015 certified; Registration # PAK17.1724-U; NTN # 0299739-8, Karachi, Pakistan
  Interventions: Drug: Allium Sativum Oil

INTERVENTIONS:
Drug: Formocresol — Formocresol will be used as non-vital pulpotomy medicament (which is gold standard)
  Other Names: medicament for Non-vital pulpotomy procedure
  Arms: Formocresol (Control-Gold standard-Group A)
Drug: Allium Sativum Oil — Allium sativum oil will be used as non-vital pulpotomy medicament compared with Formocresol (which is gold standard)
  Other Names: medicament for Non-vital pulpotomy procedure
  Arms: Allium sativum oil (Experimental-Group B)

SUMMARY:
The purpose of this randomized controlled clinical trial is to use Allium sativum oil as non-vital Pulpotomy medicament compared to Formocresol in primary teeth by evaluating its antibacterial effect against Streptococcus mutans and Lactobacillus acidophilus. It is hypothesized that there is no difference in the antibacterial effect of Allium sativum oil compared with Formocresol, when used as non-vital Pulpotomy medicaments.

DETAILED DESCRIPTION:
It is a multi-arm parallel Randomized Controlled Trial in which forty patients aged between 4 to 8 years, each containing at-least one non-vital primary molar, will be selected and randomly divided into Group A (Formocresol) and Group B (Allium sativum oil). Non-vital Pulpotomy will be performed by removing the coronal necrotic pulp. Sterile paper point will be dipped in the root canals and taken to the laboratory. Cotton pellets soaked in the respective medicaments will be placed over the root canal orifices and filled temporarily. Patients will be recalled after one week. Samples will be again taken, and tooth restored. Comparison between bacterial count at baseline and after one week of treatment will be made and expressed as Colony-Forming Units/ml (CFU/ml).

ELIGIBILITY:
Inclusion Criteria:

1. Cooperation of patients and consent of parents.
2. Patients with ASA classification I and II (mild to moderate systemic disease).
3. Non-traumatic extensively carious hence restorable primary molars.
4. No history of antibiotic use for 2 weeks.
5. Presence of following clinical signs or symptoms suggestive of non-vital tooth such as tenderness on percussion, non-responsive to cold test, periapical/furcal radiolucency, localized gingival/mucosal soreness/redness/swelling, and/or slight mobility-grade I.

Exclusion Criteria:

1. History of allergy to anesthetics and latex.
2. Radiographic evidence of pulpal floor opening into the furcation area.
3. More than half of the roots resorbed.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Antibacterial effect | 1 week
  Bacterial count of S. mutans and L. acidophilus counted as Colony Forming Units/ml (CFU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Naz, BDS, MDS, Principal Investigator — Assistant professor operative dentistry de, Montmorency College of Dentistry
Locations (1):
- de' Montmorency College of dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No